CLINICAL TRIAL: NCT04758507
Title: Targeting Gut Microbiota to Improve Efficacy of Immune Checkpoint Inhibitors in Patients With Advanced Renal Cell Carcinoma
Brief Title: Fecal Microbiota Transplantation to Improve Efficacy of Immune Checkpoint Inhibitors in Renal Cell Carcinoma
Acronym: TACITO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Dr, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2664
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To mask treatments to physicisans and recipients, both FMT bottles and syringes will be covered with dark-coloured paper before the infusion, and the patients will be unable to see the endoscopic display during the procedure. Moreover, the physicians who will evsaluate patients at follow-up will not aware of the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donor FMT (Experimental): Patients enrolled in this arm will receive donor FMT
  Interventions: Biological: donor FMT
- Placebo FMT (Placebo Comparator): Patients enrolled in this arm will receive placebo FMT (that will be made of saline solution)
  Interventions: Other: Placebo FMT

INTERVENTIONS:
Biological: donor FMT — This intervention is represented by the administration, in the recipients' gut, of donor microbiota through FMT
  Arms: Donor FMT
Other: Placebo FMT — This intervention is represented by the administration, in the recipients' gut, of a placebo through FMT
  Arms: Placebo FMT

SUMMARY:
Renal cell carcinoma (RCC) is the sixth most common cancer in men and the eighth in women in the USA. In Italy RCC incidence was 11500 new cases in 2017, while mortality was 3371 cases in 2015. Increasing evidence suggests that response to immune checkpoint inhibitors (ICIs), a novel treatment for advanced RCC (aRCC) and other epithelial tumors, can be influenced by the patient gut microbiota. Fecal microbiota transplantation (FMT) is a novel therapeutic option based on the restoration of healthy gut microbiota, and is the most effective therapy for recurrent C. difficile infection, and preliminary nonrandomized findings show that FMT is able to improve efficacy of ICIs in patients with advanced melanoma. The aim of this study is to evaluate, through a randomized controlled trial, the efficacy of targeted FMT (from donors who are responding to ICI. in improving response rates to ICIs in subjects with aRCC.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is the sixth most common cancer in men and the eighth in women in the USA. In Italy RCC incidence was 11500 new cases in 2017, while mortality was 3371 cases in 2015. Increasing evidence suggests that response to immune checkpoint inhibitors (ICIs), a novel treatment for advanced RCC (aRCC) and other epithelial tumors, can be influenced by the patient gut microbiota. Fecal microbiota transplantation (FMT) is a novel therapeutic option based on the restoration of healthy gut microbiota, and is the most effective therapy for recurrent C. difficile infection, and preliminary nonrandomized findings show that FMT is able to improve efficacy of ICIs in patients with advanced melanoma. The aim of the study is to evaluate, through a randomized controlled trial, the efficacy of targeted FMT (from donors who are responding to ICI) in improving response rates to ICIs in subjects with aRCC. So, the investigators will investigate, through a randomized controlled trial, if donor FMT will be more effective than placebo FMT in improving response to ICIs in patients with renal cell carcinoma. Patients will undergo the first infusion by colonoscopy. Then, patients will receive frozen fecal capsules (8 capsules t.i.d.) at 3 and 6 months after the first FMT.

Fifty patients will be enrolled. Sample size calculation was based on the hypothesis of the superiority of FMT+SOC over SOC alone. The 1-year PFS rate for SOC has been reported to be nearly 60%. The alternative hypothesis is that FMT can improve the 1-year PFS rate from 60% to 80% wen associated to SOC. A total of 50 patients will enter this two-treatment parallel-design study. The probability is 80 percent that the study will detect a treatment difference at a one-sided 5.0 percent significance level, if the true hazard ratio is 0.436. This is based on the assumption that the accrual period will be 36 months and the follow up period will be 36 months and the median survival is 15.1 months. The total number of events will be 37.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aRCC
* Metastatic disease (measurable and not-measurable)
* Radiological assessment within 8 wks before enrollment
* Patient eligible to therapy with ICI for aRCC (or started within 8 wks)
* Ability to provide written informed consent
* Ability to be compliant with the scheduled procedures

Exclusion Criteria:

* Major comorbidities
* Concomitant GI or autoimmune disorders, or HIV, HBV, HCV infection
* Continuative corticosteroid therapy
* Previous treatment with systemic immune-suppressants or immune-modulatory drugs
* Antibiotic therapy within 4 weeks prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Number of participants who will be free from tumor progression, as assessed by RECIST criteria v. 1.1. | 12 months
  The investigators will evaluate the number of participants who will be free from tumor progression, as assessed by RECIST criteria v. 1.1., after treatments, at 12 month-follow-up

SECONDARY OUTCOMES:
Number of participants who will obtain a partial or a complete tumor response to immunotherapy, as assessed by RECIST criteria v. 1.1, after treatments | 12 months
  The investigators will evaluate the number of participants who will obtain a partial or a complete tumor response to immunotherapy, as assessed by RECIST criteria v. 1.1, after treatments, at 12 month-follow-up
Number of participants who will die for any reason (overall survival) | 12 months
  The investigators will evaluate the number of participants who will die for any reason throughout the study period (12 months)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  The number of participants with treatment-related adverse events (assessed by CTCAE v4.0) will be recorded throughout the study period (12 months)
Number of participants with significant increase in alpha-diversity (assessed by Shannon index) and beta-diversity (assessed by Bray-Curtis dissimilarity) of their gut microbiota after treatments | 12 months
  Throughout the study period (12 months) the investigators will evaluate the number of participants with significant increase in alpha-diversity (assessed by Shannon index) and beta-diversity (assessed by Bray-Curtis dissimilarity) of their gut microbiota after treatments, compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ianiro, MD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (2):
- Italy (2):
  - Digestive Disease Center, Rome, Rome
  - Gianluca Ianiro, Rome, Rome

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon request to the PI

REFERENCES:
- [Background] Ianiro G, Rossi E, Thomas AM, Schinzari G, Masucci L, Quaranta G, Settanni CR, Lopetuso LR, Armanini F, Blanco-Miguez A, Asnicar F, Consolandi C, Iacovelli R, Sanguinetti M, Tortora G, Gasbarrini A, Segata N, Cammarota G. Faecal microbiota transplantation for the treatment of diarrhoea induced by tyrosine-kinase inhibitors in patients with metastatic renal cell carcinoma. Nat Commun. 2020 Aug 28;11(1):4333. doi: 10.1038/s41467-020-18127-y. PMID 32859933
- [Background] Baruch EN, Youngster I, Ben-Betzalel G, Ortenberg R, Lahat A, Katz L, Adler K, Dick-Necula D, Raskin S, Bloch N, Rotin D, Anafi L, Avivi C, Melnichenko J, Steinberg-Silman Y, Mamtani R, Harati H, Asher N, Shapira-Frommer R, Brosh-Nissimov T, Eshet Y, Ben-Simon S, Ziv O, Khan MAW, Amit M, Ajami NJ, Barshack I, Schachter J, Wargo JA, Koren O, Markel G, Boursi B. Fecal microbiota transplant promotes response in immunotherapy-refractory melanoma patients. Science. 2021 Feb 5;371(6529):602-609. doi: 10.1126/science.abb5920. Epub 2020 Dec 10. PMID 33303685
- [Background] Davar D, Dzutsev AK, McCulloch JA, Rodrigues RR, Chauvin JM, Morrison RM, Deblasio RN, Menna C, Ding Q, Pagliano O, Zidi B, Zhang S, Badger JH, Vetizou M, Cole AM, Fernandes MR, Prescott S, Costa RGF, Balaji AK, Morgun A, Vujkovic-Cvijin I, Wang H, Borhani AA, Schwartz MB, Dubner HM, Ernst SJ, Rose A, Najjar YG, Belkaid Y, Kirkwood JM, Trinchieri G, Zarour HM. Fecal microbiota transplant overcomes resistance to anti-PD-1 therapy in melanoma patients. Science. 2021 Feb 5;371(6529):595-602. doi: 10.1126/science.abf3363. PMID 33542131
- [Background] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Derived] Porcari S, Ciccarese C, Heidrich V, Rondinella D, Quaranta G, Severino A, Arduini D, Buti S, Fornarini G, Primi F, Stumbo L, Giannarelli D, Giudice GC, Damassi A, Giron Berrios JR, Puncochar M, Barbazuk TB, Piccinno G, Pinto F, Armanini F, Asnicar F, Schinzari G, Derosa L, Kroemer G, Sanguinetti M, Masucci L, Gasbarrini A, Tortora G, Cammarota G, Zitvogel L, Segata N, Iacovelli R, Ianiro G. Fecal microbiota transplantation plus pembrolizumab and axitinib in metastatic renal cell carcinoma: the randomized phase 2 TACITO trial. Nat Med. 2026 Jan 28. doi: 10.1038/s41591-025-04189-2. Online ahead of print. PMID 41606119